CLINICAL TRIAL: NCT04557267
Title: Dose-ranging Study of Labisia Pumila Aqueous Ethanolic Standardized Extract (SKF7™) for Obesity: a Randomized, Double-blind, Placebo-controlled, Phase-2 Study
Brief Title: Dose-ranging Study of SKF7™ for Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Medika Natura Sdn Bhd (Industry)
Responsible Party: Principal Investigator, Nafrialdi, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CRSU.P.SKF7F2/1019/04.08
Record Dates: First submitted 2020-09-07; First posted 2020-09-21 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Obesity
Keywords: dose-ranging; Kacip Fatimah; Labisia pumila; obesity
MeSH Terms: conditions — Obesity | interventions — Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: 4 parallel groups, 3 doses of study drug versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active drug and placebo are made in similar
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (dosage A) (Experimental): The lower dose of the active drug
  Interventions: Drug: low-dose
- Group B (dosage 2) (Experimental): The middle dose of the active drug
  Interventions: Drug: Middle-dose
- Group C (dosage 3) (Experimental): The higher dose of the active drug
  Interventions: Drug: Higher-dose
- Group D (placebo) (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: low-dose — Dosage 1
  Arms: Group A (dosage A)
Drug: Middle-dose — Dosage 2
  Arms: Group B (dosage 2)
Drug: Higher-dose — Dosage 3
  Arms: Group C (dosage 3)
Drug: Placebo — Placebo
  Arms: Group D (placebo)

SUMMARY:
This study has been designed as a randomized, double blinded, multi-centric, placebo controlled, and phase II dose-ranging study. The herbal drug contains bioactive ingredients from Labisia pumila plant and it is an aqueous ethanolic standardized extract (SKF7™).

DETAILED DESCRIPTION:
Labisia pumila or Kacip Fatimah is a native Malaysian and Indonesian plant. It has been used as traditional medicine for over 400 years by both men and women for multiple treatments including toning and firming the abdominal area. As a water-ethanol dry extract, it has been reported to reduce body weight, cholesterol level and triglyceride level, and regulate blood glucose and sex hormones. In Malaysia, this Kacip Fatimah extract has been used as a natural anti-obesity drug and dietary supplement for healthy weight loss and healthy body by the trade-name of Labeesity® or SKF7™. This extract has been shown to be pesticide / herbicide free and has branded halal ingredient identity and security.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18 - 50 yrs or women aged 18 until before perimenopause, with obesity
2. Willing to participate in the study by signing the informed consent
3. Healthy by anamnesis
4. Agreed to maintain their current lifestyles (no changes in their diet and physical exercise) during the clinical trial period.

Exclusion Criteria:

1. Positive result for Rapid test for COVID-19 at screening period.
2. Known hypersensitivity to any herbal product.
3. Pregnant or lactating women.
4. Taking any other weight loss therapy and/or lipid lowering products.
5. Participate in other interventional clinical study or have taken other investigational drug within 30 days prior to screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-22 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 12 weeks
  Percentage of subjects whose Body Weight is lowered
Change in waist and hip circumferences | 12 weeks
  Change in waist and hip circumference
Change in the waist-hip and waist-height ratios | 12 weeks
  Change in waist-hip ratio and waist-height ratio
Change in Body Mass Index (BMI) | 12 weeks
  Change in BMI in kg/m^2

SECONDARY OUTCOMES:
Body fat percentage | 12 weeks
  The change of body fat percentage
Lean Body Mass | 12 weeks
  The amount of lean body mass will be calculated from body fat percentage

OTHER OUTCOMES:
Incidence of abnormal vital signs and of abnormal laboratory test results | 12 weeks
  Abnormality of vital signs and laboratory test results
Incidence of Adverse Events | 12 weeks
  The incidence and percentage of Adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Arini Setiawati, PhD, Study Chair — Clinical Research Supporting Unit, Faculty of Medicine, University of Indonesia; Nafrialdi Agus, MD, PhD, Principal Investigator — Pharmacology & Therapeutics, Faculty of Medicine, Universitas Indonesia
Locations (3):
- Indonesia (3):
  - Indonesia Medical Education and Research Institute, Jakarta, DKI Jakarta
  - Faculty of Medicine, Krida Wacana Christian University, Jakarta, DKI Jakarta
  - Makara Satellite Clinic, Depok, West Java

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee S, Lee H, Cho Y, Kim J, Kang JW, Seo BK, Baek YH, Lee JD. The efficacy and safety of Hanslim for obese patients: Study protocol for a multicenter, randomized, double-blind, multi-dose, placebo-controlled, phase IIb clinical trial. Medicine (Baltimore). 2018 Sep;97(38):e12440. doi: 10.1097/MD.0000000000012440. PMID 30235727
- See also: EMA Guideline on clinical evaluation of medicinal products used in weight control — https://www.ema.europa.eu/en/documents/scientific-guideline/guideline-clinical-evaluation-medicinal-products-used-weight-management-revision-1_en.pdf
- See also: The Asia-Pacific Perspective: Redefining Obesity and its Treatment — https://apps.who.int/iris/handle/10665/206936